CLINICAL TRIAL: NCT02171468
Title: Pharmacokinetics, Safety and Pharmacodynamics After Multiple Oral Doses of Dabigatran Etexilate Capsule (110 mg and 150 mg b.i.d., 7 Days) in Healthy Japanese and Caucasian Male Subjects (Open Label Study)
Brief Title: Pharmacokinetics, Safety and Pharmacodynamics After Multiple Oral Doses of Dabigatran Etexilate Capsule in Healthy Japanese and Caucasian Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.61
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (2):
- Dabigatran high dose (Experimental)
  Interventions: Drug: Dabigatran high dose
- Dabigatran low dose (Experimental)
  Interventions: Drug: Dabigatran low dose

INTERVENTIONS:
Drug: Dabigatran high dose
  Arms: Dabigatran high dose
Drug: Dabigatran low dose
  Arms: Dabigatran low dose

SUMMARY:
To investigate and compare pharmacokinetics, safety and pharmacodynamics of dabigatran etexilate following oral administration of multiple doses (110 mg and 150 mg b.i.d., 7 days) in healthy male subjects between Japanese and Caucasians

ELIGIBILITY:
Inclusion Criteria:

1. Japanese or Caucasian healthy male subjects according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate and body temperature), 12-lead electrocardiogram, clinical laboratory tests
   * No finding of clinical relevance
   * No evidence of a clinically relevant concomitant disease
   * Caucasian subjects are from a well-defined Caucasian population, both parents of Caucasians, the subjects can understand the subject information for informed consent in English and the subjects have lived 8 or less than 8 years in Japan
2. Age: ≥20 and ≤45 years
3. Body mass index (BMI): ≥18.5 and ≤29.9 kg/m2
4. Signed and dated written informed consent before admission to the trial site

Exclusion Criteria:

1. Current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Subject can not use an adequate form of contraception from the time of the first dose on Day 1 up to end-of study examination
3. Current diseases of the central nervous system (such as epilepsy), or psychiatric disorders or neurological disorders
4. History of clinically significant orthostatic hypotension, clinically significant current or past fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of

   * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the safety assessment as judged by the investigator (excluding asymptomatic seasonal rhinitis/hay fever)
   * any bleeding disorder including prolonged or habitual bleeding
   * other hematologic diseases
   * cerebral bleeding (e.g. after a car accident)
   * concussions (head trauma resulting in injuring to brain) with or without loss of consciousness
7. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives, whichever is shorter, of the respective drug prior to administration or during the trial
8. Use of aspirin (including over-the-counter medications), antipletelet agents like ticlopidine or dipyridamole, chronic administration of nonsteroidal antiinflammatory drugs , coumadin like anticoagulants, chronic use of corticosteroids, heparin or fibrinolytic agents within 28 days prior to administration up to end-of-study examination
9. Participation in another trial with an investigational drug within 3 months prior to administration up to end-of-study examination
10. Smoker (>10 cigarettes/day or inability to refrain from smoking during the trial)
11. Alcohol abuse (more than 60 g/day; confirmed by interview)
12. Drug abuse (confirmed by interview)
13. Blood donation (more than 100 mL from 3 months prior to screening and any blood donation from screening up to end-of-study examination)
14. Excessive physical activities (within 7 days prior to the first drug administration up to end-of-study examination)
15. Any laboratory value outside the reference range that is of clinical relevance
16. Known hypersensitivity to the investigational drug or its excipients
17. Subject who was judged ineligible by the investigator or the sub-investigator
18. History of any familial bleeding disorder
19. Thrombocytes <15 x 10**4 /microL

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | up to 10 days
Changes in QT(c) intervals | up to 7 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state) | up to 7 days
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 7 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration) | day 1
tmax (time from dosing to maximum measured concentration) | day 1
AUCτ,1 (area under the concentration-time curve over a uniform dosing interval τ after administration of single dose on Day 1) | day 1
tmax,ss (time from last dosing to maximum concentration at steady state) | up to 7 days
Cmin,ss (minimum concentration at steady state over a uniform dosing interval τ) | up to 7 days
λz,ss (terminal rate constant at steady state) | up to 7 days
t1/2,ss (terminal half-life at steady state) | up to 7 days
MRTpo,ss (mean residence time in the body at steady state after oral administration) | up to 7 days
CL/F,ss (apparent clearance in the plasma at steady state after extravascular multiple dose administration) | up to 7 days
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 7 days
RA,Cmax,13 (accumulation ratio calculated as Cmax,ss/Cmax) | up to 7 days
RA,AUC,13 (accumulation ratio calculated as AUCτ,ss/AUCτ,1) | up to 7 days
area under the curve for activated partial thromboplastin time (aPTT) | 0 - 12 hours after adminstration on day 1 and day 7
area under the curve for ecarin clotting time (ECT) | 0 - 12 hours after adminstration on day 1 and day 7
comparison of trough concentrations | after doses 3, 5, 7, 9, 11 and 13
comparison of trough concentrations morning versus evening | after doses 9, 10, 11, 12, 13